CLINICAL TRIAL: NCT06660524
Title: Clinical Study on the Influence of Calcium and Phosphorus Regulation Therapy on Valvular Heart Disease.
Brief Title: Calcium-Phosphorus Regulation Therapy on Heart Valve Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-GSP-GG-38
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Degenerative Heart Valve Disease; Heart Valve Calcification; Chronic Kidney Disease(CKD); Calcium-Phosphorus Metabolism Disorders
Keywords: Heart Valve Calcification; Degenerative Valve Disease; Chronic Kidney Disease; Calcium-Phosphorus Regulation; Sevelamer
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer; Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Randomized grouping is generated by applying the data entry platform. According to the randomization results, the experimental group is given a sevelamer prescription, and the control group is given a calcium carbonate prescription.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sevelamer Treatment (Experimental): Sevelamer is administered orally, and the administration strategy is implemented in accordance with the 2017 KDIGO Guideline and the 2019 Chinese Guideline for the Diagnosis and Treatment of Mineral and Bone Disorders in Chronic Kidney Disease.
  Interventions: Drug: Sevelamer
- Calcium Carbonate Treatment (Active Comparator): Calcium carbonate is administered orally, and the administration strategy is implemented in accordance with the 2017 KDIGO Guideline and the 2019 Chinese Guideline for the Diagnosis and Treatment of Mineral and Bone Disorders in Chronic Kidney Disease.
  Interventions: Drug: Calcium carbonate

INTERVENTIONS:
Drug: Sevelamer — Sevelamer is administered orally, and the administration strategy is implemented in accordance with the 2017 KDIGO Guideline and the 2019 Chinese Guidelines for the Diagnosis and Treatment of Mineral and Bone Disorders in Chronic Kidney Disease.
  Arms: Sevelamer Treatment
Drug: Calcium carbonate — Calcium carbonate is administered orally, and the administration strategy is implemented in accordance with the 2017 KDIGO Guideline and the 2019 Chinese Guideline for the Diagnosis and Treatment of Mineral and Bone Disorders in Chronic Kidney Disease.
  Arms: Calcium Carbonate Treatment

SUMMARY:
The goal of this clinical trial is to learn if calcium-phosphorus regulation therapy can slow the progression of heart valve calcification in patients with degenerative heart valve disease and chronic kidney disease (CKD). The main questions it aims to answer are:

* Does Sevelamer lower the progression of heart valve calcification compared to calcium carbonate over 12 months?
* What are the impacts of calcium-phosphorus regulation therapy on major cardiovascular events such as heart failure, cardiovascular death, and the need for valve surgery? Researchers will compare Sevelamer to calcium carbonate to see if Sevelamer is more effective in reducing heart valve calcification.

Participants will:

* Take Sevelamer or calcium carbonate daily for 12 months.
* Undergo echocardiography and CT scans at baseline and after 12 months to assess heart valve calcification.
* Attend follow-up visits at 3, 6, 9, and 12 months to monitor blood tests and adjust treatment as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old.

  * Degenerative valvular heart disease clearly diagnosed by ultrasound or clinical history with calcification manifestation (including no stenosis or insufficiency due to calcification, mild, moderate and severe stenosis and insufficiency caused by calcification).

    * Glomerular filtration rate < 60 mL/min (CKD-EPI formula).

      * Serum phosphorus > 1.45 mmol/L (4.5 mg/dl).

Exclusion Criteria:

* Patients refuse to sign the informed consent form for the study.

  * Non-degenerative valvular heart disease even if there is valvular calcification, such as rheumatic valvular heart disease, congenital valvular heart disease, etc.

    * Valve lesions are evaluated by cardiac surgeons and have indications for surgical thoracotomy or interventional medical treatment and there are no surgical contraindications.

      * Life expectancy less than 1 year. ⑤ Abnormal parathyroid function.

        * Those with renal insufficiency who are planned to undergo dialysis treatment within half a year.

          * Malignant tumor.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The change of valve calcification score on CT scan from baseline to 1 year of treatment. | from baseline to 1 year of treatment
  The change of valve calcification score on CT scan from baseline to 1 year of treatment.

SECONDARY OUTCOMES:
major cardiovascular events | from baseline to 1 year of treatment
  The composite endpoint of major cardiovascular events includes hospitalization or outpatient/emergency department visits due to heart failure; cardiovascular death; undergoing interventional/surgical valve surgery; and non-fatal myocardial infarction.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Doris MK, Jenkins W, Robson P, Pawade T, Andrews JP, Bing R, Cartlidge T, Shah A, Pickering A, Williams MC, Fayad ZA, White A, van Beek EJ, Newby DE, Dweck MR. Computed tomography aortic valve calcium scoring for the assessment of aortic stenosis progression. Heart. 2020 Dec;106(24):1906-1913. doi: 10.1136/heartjnl-2020-317125. Epub 2020 Oct 5. PMID 33020228
- [Background] Williams MC, Massera D, Moss AJ, Bing R, Bularga A, Adamson PD, Hunter A, Alam S, Shah ASV, Pawade T, Roditi G, van Beek EJR, Nicol ED, Newby DE, Dweck MR. Prevalence and clinical implications of valvular calcification on coronary computed tomography angiography. Eur Heart J Cardiovasc Imaging. 2021 Feb 22;22(3):262-270. doi: 10.1093/ehjci/jeaa263. PMID 33306104
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Meng Z, Li Z, Zhang E, Zhang L, Liu Q, Wu Y. Sevelamer Attenuates Bioprosthetic Heart Valve Calcification. Front Cardiovasc Med. 2021 Sep 29;8:740038. doi: 10.3389/fcvm.2021.740038. eCollection 2021. PMID 34660741
- [Background] Hoevelmann J, Mahfoud F, Lauder L, Scheller B, Bohm M, Ewen S. Valvular heart disease in patients with chronic kidney disease. Herz. 2021 Jun;46(3):228-233. doi: 10.1007/s00059-020-05011-0. Epub 2021 Jan 4. PMID 33394059
- [Background] Urena-Torres P, D'Marco L, Raggi P, Garcia-Moll X, Brandenburg V, Mazzaferro S, Lieber A, Guirado L, Bover J. Valvular heart disease and calcification in CKD: more common than appreciated. Nephrol Dial Transplant. 2020 Dec 4;35(12):2046-2053. doi: 10.1093/ndt/gfz133. PMID 31326992
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Update Work Group. KDIGO 2017 Clinical Practice Guideline Update for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl (2011). 2017 Jul;7(1):1-59. doi: 10.1016/j.kisu.2017.04.001. Epub 2017 Jun 21. No abstract available. PMID 30675420
- [Background] Blaser MC, Kraler S, Luscher TF, Aikawa E. Multi-Omics Approaches to Define Calcific Aortic Valve Disease Pathogenesis. Circ Res. 2021 Apr 30;128(9):1371-1397. doi: 10.1161/CIRCRESAHA.120.317979. Epub 2021 Apr 29. PMID 33914608
- [Background] Rossebo AB, Pedersen TR, Boman K, Brudi P, Chambers JB, Egstrup K, Gerdts E, Gohlke-Barwolf C, Holme I, Kesaniemi YA, Malbecq W, Nienaber CA, Ray S, Skjaerpe T, Wachtell K, Willenheimer R; SEAS Investigators. Intensive lipid lowering with simvastatin and ezetimibe in aortic stenosis. N Engl J Med. 2008 Sep 25;359(13):1343-56. doi: 10.1056/NEJMoa0804602. Epub 2008 Sep 2. PMID 18765433
- [Background] Moura LM, Ramos SF, Zamorano JL, Barros IM, Azevedo LF, Rocha-Goncalves F, Rajamannan NM. Rosuvastatin affecting aortic valve endothelium to slow the progression of aortic stenosis. J Am Coll Cardiol. 2007 Feb 6;49(5):554-61. doi: 10.1016/j.jacc.2006.07.072. Epub 2007 Jan 22. PMID 17276178
- [Background] Chan KL, Teo K, Dumesnil JG, Ni A, Tam J; ASTRONOMER Investigators. Effect of Lipid lowering with rosuvastatin on progression of aortic stenosis: results of the aortic stenosis progression observation: measuring effects of rosuvastatin (ASTRONOMER) trial. Circulation. 2010 Jan 19;121(2):306-14. doi: 10.1161/CIRCULATIONAHA.109.900027. Epub 2010 Jan 4. PMID 20048204
- [Background] Yadgir S, Johnson CO, Aboyans V, Adebayo OM, Adedoyin RA, Afarideh M, Alahdab F, Alashi A, Alipour V, Arabloo J, Azari S, Barthelemy CM, Benziger CP, Berman AE, Bijani A, Carrero JJ, Carvalho F, Daryani A, Duraes AR, Esteghamati A, Farid TA, Farzadfar F, Fernandes E, Filip I, Gad MM, Hamidi S, Hay SI, Ilesanmi OS, Naghibi Irvani SS, Jurisson M, Kasaeian A, Kengne AP, Khan AR, Kisa A, Kisa S, Kolte D, Manafi N, Manafi A, Mensah GA, Mirrakhimov EM, Mohammad Y, Mokdad AH, Negoi RI, Thi Nguyen HL, Nguyen TH, Nixon MR, Otto CM, Patel S, Pilgrim T, Radfar A, Rawaf DL, Rawaf S, Rawasia WF, Rezapour A, Roever L, Saad AM, Saadatagah S, Senthilkumaran S, Sliwa K, Tesfay BE, Tran BX, Ullah I, Vaduganathan M, Vasankari TJ, Wolfe CDA, Yonemoto N, Roth GA; Global Burden of Disease Study 2017 Nonrheumatic Valve Disease Collaborators. Global, Regional, and National Burden of Calcific Aortic Valve and Degenerative Mitral Valve Diseases, 1990-2017. Circulation. 2020 May 26;141(21):1670-1680. doi: 10.1161/CIRCULATIONAHA.119.043391. Epub 2020 Mar 29. PMID 32223336